CLINICAL TRIAL: NCT03130712
Title: ￼An Open-label, Uncontrolled, Single-arm Pilot Study to Evaluate Intratumor Injection Mediated GPC3-targeted Chimeric Antigen Receptor T Cells in Advanced Hepatocellular Carcinoma
Brief Title: A Study of GPC3-targeted T Cells by Intratumor Injection for Advanced HCC (GPC3-CART)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai GeneChem Co., Ltd. (Industry)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 302 GPC3-CART
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Carcinoma, Hepatocellular
Keywords: immunotherapy; GPC3-CART; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GPC3-CART cells (Experimental)
  Interventions: Drug: GPC3-CART cells

INTERVENTIONS:
Drug: GPC3-CART cells — Intratumol injection as a local drug delivery pathway, so that more T cells gathered at the tumor site, less T cells to migrated to the normal tissue, thereby enhancing the efficacy of anti-tumor, reducing the potential of side effects. And GPC3-CART is a 2nd CAR, with GPC3 as the target protein, 4-1BB as a co- stimulator

SUMMARY:
In this study, CART cells are targeted to GPC3 by intratumor injected that we hope by this means could improve the local CAR-T cell numbers, meanwhile reduce the potential side effects.

DETAILED DESCRIPTION:
Patients treated with leukapheresis to obtain peripheral blood mononuclear cells, and then PBMC are purified. T cells are activated and then re-engineered to express chimeric antigen receptors (CARs) specific for GPC3. Cells are expanded in culture and returned to the participant by intratumor injection at the dose of(1-10)×106 CAR positive T cells. The cells perfusion process would only last for (1-2) min. GPC-CART cells are injected into each tumor focus only once.

ELIGIBILITY:
Inclusion Criteria:

* Advanced HCC patients with age between 18 and 69 years old;
* Persistent cancer after at least one prior standard of chemotherapy or surgery, and without high level evidence of second-line treatment;
* The intended intratumoral injection sites of tumor can be showed clear by CT or ultrasound scan, and safe access to without important neuromuscular pass;
* The ECOG score less than 1 points, and the expected survival more than 4 months;
* Recovery from previous treatment: all side effects (except hair loss) were reduced to level 1 or below, according to NCI-CTC AE version 4;
* Pregnancy test (urine beta -HCG) negative (for women of childbearing age);
* Meet one of the following conditions:

  1. GPC3 was expressed in more than 15% of tumor cells (immunohistochemical method)
  2. GPC3 expression in more than 30% of tumor cells (flow cytometry);
* Satisfactory organ and bone marrow function as defined by the following: (1) creatinine <1.5mg/dl; (2) albumin >2; (3) cardiac ejection fraction of >55%; (4) hemoglobin>9g/dl, bilirubin 2.0×the institution normal upper limit;
* Adequate venous access for apheresis;
* Voluntary informed consent.

Exclusion Criteria:

* Pregnant or lactating women, urine pregnancy test was positive before transplantation of CAR-T cells 48 hours;
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary;
* Patients in the situation of: (1) 30 days before apheresis is still in the period of other antitumor drug observation; (2) patient dont recuperate from earlier acute adverse influence brought by any treatments accepted before;
* Four weeks before recruit accepted radiation therapy; Previously treatment with any gene therapy products;
* Feasibility assessment during screening demonstrates<30% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation;
* Any serious, uncontrolled diseases (including, but not limit to, unstable angina pectoris, congestive heart failure, grade III or IV cardiac disease, serious arrhythmia, liver and kidney disorders or metabolic diseases, CNS diseases);
* Patient with severe acute hypersensitive reaction;
* Forced position, can not be adjusted according to requirements;
* Severe heart, lung, liver, kidney function, blood coagulation dysfunction;
* Taking part in other clinical trials;
* Study leader considers not suitable for this tiral.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety of CAR-T cell infusion mediated by intratumoral injection as measured by number of participants with adverse Events | 6 weeks
  To determine the safety and regimen limiting toxicity (RLT) of anti-GPC3 CAR-T intratumoral injection for GPC3-expressing HCC.

SECONDARY OUTCOMES:
Number of participants with tumor response as measured by RECIST | 8 weeks]
Serum cytokine levels | 8 weeks
  Measurement of cytokines as indicators of immune response, including IL-2/IL-6/IL-10/TNF/IL-2R

CONTACTS AND LOCATIONS:
Overall Officials: Lu Yinying, Doctor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- 302 Military Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided